CLINICAL TRIAL: NCT02506725
Title: Quarenta Semanas: Innovative Intervention in Prenatal Care for Reduction of Prematurity
Acronym: quarenta
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oswaldo Cruz Foundation (Other)
Collaborators: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Maria Elisabeth Lopes Moreira, MD,PHD, Oswaldo Cruz Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OswaldoCruz
Record Dates: First submitted 2015-07-20; First posted 2015-07-23 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Pregnancy
Keywords: prenatal care; pregnancy; prematurity
MeSH Terms: conditions — Premature Birth | interventions — Prenatal Care; Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: statistician and qualitative researchers
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prenatal Care in groups (Experimental): We will do prenatal care using centering care pregnancy methodology in 10 sessions
  Interventions: Other: prenatal care in groups
- Control Group (No Intervention): We will do in this arm conventional Prenatal care available in the family clinics

INTERVENTIONS:
Other: prenatal care in groups — We will do prenatal care in groups using centering care pregnancy methodology
  Other Names: centering care for prenatal
  Arms: Prenatal Care in groups

SUMMARY:
The goal of Quarenta Semanas is to remove risk factors for preterm birth by linking women to prenatal care in the first trimester; supporting, educating and empowering women in pregnancy to reduce maternal stress and interrupt social, psychological, attitudinal and biological risk factors for preterm birth; and providing evidence-based, quality care that identifies and intervenes medically to treat underlying chronic and emergent conditions associated with preterm birth.

DETAILED DESCRIPTION:
Brazil is among 10 countries with the highest rates of preterm birth (12.4%). Alarmingly, rates are rising. Research has identified multiple risk factors for preterm birth, which can be grouped into four domains, all of which must be addressed to result in meaningful reductions in preterm birth. Domain 1: Access to and utilization of prenatal care. With universal access to prenatal and postpartum care assured via Brazil's Stork Network, Community Health Workers will conduct neighborhood outreach to identify women early in pregnancy and assure that women use prenatal services in the first trimester.

Domain 2: Maternal social, demographic and attitudinal risk factors include maternal stress, lack on knowledge about pregnancy, lack of social support, feeling low control over their health and pregnancy care, unplanned or unwanted pregnancy, unsatisfactory relationship with the father, social isolation, and short interpregnancy interval. Maternal demographic characteristics (e.g., Black race, being single, maternal age under 21 or over 35 years, and poverty) are helpful for identifying high-risk women, but are less amenable to interventions to prevent preterm birth. Domain 3: Maternal physical health risk factors include prior preterm birth, multiple gestation, infection, mucosal or systemic immune responses, diabetes, under and overweight, and hypertension. Several of these factors may be prevented or treated with optimal medical care. Domain 4: Quality of prenatal care includes completing all prenatal care visits, provider compliance with prenatal care guidelines, access to recommended tests or equipment, and appropriate referral of high-risk pregnant women to specialty care. QS is designed to attenuate the effects of risk factors for preterm births in each of these four domains through early access to high quality prenatal care delivered in a group model. STUDY DESIGN The Randomized Trial Framework. We will implement QS in the context of a RCT. We recruited 4 clinics in the Stork Network that serve the same patient population and geographic area in the central and west area of Rio de Janeiro. We will pair them into 2 dyads matched by number of prenatal patients served. We will randomly assign one clinic in each dyad to implement QS and the other will continue to deliver care as usual. Below, when we describe activities related to QS, they will be done only in the 2 QS clinics; in the control clinics, we will collect data only. The clinics or Health Municipal Centers belong to the Municipal Health System. They are staffed by Family Doctors, Nurses and Health Agents and look after a specific geographic location. They provide prenatal care and are able to perform laboratory tests, X-rays and obstetrical ultrasonography. Clinics selected for this project follow at least 250 pregnant women per year. The 2 QS sites are intervention sites and two are control sites. All sites have WiFi or wired internet access for REDCap survey administration, which is web based. The targeted enrollment is 240 QS women, 20 groups of 12 women. In each of the two QS clinical sites, we will form one group per month for 10 months, totaling 20 groups. We will enroll an equivalent number of women in the control clinics matching the pace of recruitment in the QS clinics. We will track that the appropriate number of groups are started and that the meetings occur monthly from 16-32 weeks and then biweekly thereafter until delivery. The "Centering Care Pregnancy" methodology will be used in the intervention clinics in prenatal care in groups.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study:

* women must be at least eighteen years old and pregnant.
* They must be less than 12 weeks pregnant at the time of enrollment.
* They must speak Portuguese.
* Multiple gestation pregnancies will be excluded.

Exclusion Criteria:

* women who submit reasons not to take part groups after applying the questionnaire

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
prematurity rate | 12 months
  birth before 37 weeks of gestational age

SECONDARY OUTCOMES:
mothers satisfaction | 12 months
  scale to do measurement of mothers satisfaction
vaginal birth | 12 months
  % of normal birth

CONTACTS AND LOCATIONS:
Overall Officials: Shioban Dolan, MD, Study Director — Montefiore Medical Center
Locations (1):
- Maria Elisabeth Moreira, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No